CLINICAL TRIAL: NCT04533126
Title: Canaux de COmmuniCAtion et Fonctionnement du CErveau: Étude Pilote en IRMf
Brief Title: Channels of Communication & Brain Functioning: Pilot fMRI Study
Acronym: COCACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: Kahler Communication France (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHAO20-WEH-COCACE (DR200102)
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Communication; Personality
Keywords: Communication channel; Personality; Brain network; fMRI; Process communication model
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Communication is a social process involving individuals exchanging messages. It is usual to observe different reactions according to the manner of communication, the manner in which such information is exchanged.

In this work, it will be examined how different communication modalities cause different reactions in a person. We make the assumption that each communication modality is based on a different brain network.

DETAILED DESCRIPTION:
This work will use the Process Communication Model (PCM) that is a tool based on human behavior, created by Taibi Kahler. It helps to understand how people interact and communicate. In order to communicate well with a person, it is convenient to use an adapted channel of communication. PCM focuses on the mastery of fundamental communication skills that are required to adapt and connect with all types of people. The sets of adaptive communications skills are learning, assessing, adapting, predicting and resolution. PCM defines six basic personality types, and four different channels of communication. Each one has one or several favourite channels of communication. On the whole, there are the following four channels of communication: Prescriptive, Informative-Interrogative, fostering, Emotional-Ludic.

* In the prescriptive channel, the interlocutor should be firm and determined, without being aggressive.
* The informative/interrogative channel requires a neutral tone of voice, showing no particular emotion. The interlocutor should emphasize using questions as a tool to communicate with the person.
* The ludic/emotive channel emphasizes exclamations, interjections, and allows expressing one's desires and urges, with immediate reactions without thinking them twice.
* The fostering channel allows sharing one's emotions and feelings with the interlocutor in a close, warm, and caring way.

These channels refer to both the used words and to the non-verbal part of communication (gestures, mimic, tone of voice).

This study aims to characterize the brain regions involved in the response to the different channels of communication.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers.
2. Both sexes (1:1).
3. Aged between 20 and 30 years old.
4. Medical student, from L2.
5. A person who has signed a written, free and informed consent.
6. Person affiliated to a social security scheme.

Exclusion Criteria:

1. Current clinically significant psychiatric disorder (MINI 7.0): mood disorder, bipolar disorder, psychotic disorder, substance abuse.
2. Current or past neurological disorder with current functional impact.
3. Chronic unstable somatic pathology.
4. Occasional use of medication other than contraceptives, migraine medication, or analgesics.
5. MRI contraindications, including claustrophobia.
6. Pregnant or breastfeeding woman.
7. Subject deprived of liberty (by a judicial or administrative decision).
8. Subject protected by law (subject under guardianship and curatorship).
9. Legal incapacity and/or other circumstances rendering the subject incapable of understanding the nature, purpose or consequences of the study.
10. A person participating in a clinical drug study or in a period of exclusion from any clinical study due to previous participation.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants, medical students
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes in fMRI activity level | 1-day
  Measure the differences in fMRI BOLD activation in healthy subjects while viewing typical videos of four different types of communication channels.

CONTACTS AND LOCATIONS:
Overall Officials: GISSOT Valérie, MD, Principal Investigator — CHRU Tours - CIC1415
Locations (1):
- Centre Investigation Clinique, Tours, Centre-Val de Loire, France

IPD SHARING:
Plan to Share IPD: No